CLINICAL TRIAL: NCT01065896
Title: The Use of Non-invasive Multidetector Coronary Computed Tomography Imaging for the Assessment of Coronary Calcification in Persons With Spinal Cord Injury
Brief Title: Coronary Computed Tomography (CT) to Measure Coronary Calcification in Spinal Cord Injury (SCI)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-12
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; coronary artery disease
MeSH Terms: conditions — Spinal Cord Injuries; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Although conventional risk factors for coronary heart disease (CHD) have been identified and routinely used to determine risk for CHD in the general population, a systematic approach to determine population-specific risk for CHD has not been performed prospectively in those with SCI. CHD is a leading cause of death in spinal cord injury, occurring at younger ages than in the able-bodied population. Conventional risk factors for CHD are high serum concentrations of low-density lipoprotein (LDL), low serum concentrations of high-density lipoprotein (HDL), diabetes mellitus (DM), positive smoking history, and positive family history of premature CHD.

Coronary calcification (CAC) is a commonly occurring phenomenon that does not necessarily indicate significant obstructive disease. Studies have shown that a strong association exists between coronary calcification and coronary heart disease. The purpose of this study is to compare the CAC scores in persons with SCI with a historical control group of able-bodied persons from a national data base who will be matched for conventional risk factors for coronary artery disease (CAD) and to determine the relationship between CAC scores and conventional and emerging risk factors for CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age;
2. Chronic (e.g., duration of injury at least 6 months), stable SCI (regardless of level of lesion or completeness of injury);
3. Concurrently participating in or previously completed protocol # 0454-06-073, "Risk Factors for Coronary Heart Disease in Spinal Cord Injury: conventional and emerging".

Exclusion Criteria:

1. Acute medical illness;
2. Pregnancy (as determined by a pregnancy test < 1 week of the study); and
3. The presence of a chronic disease (i.e., heart disease, pulmonary disease, etc.);
4. Inability to comply with breathing instructions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCI subjects will be included in the study if they have moderate or high risk for coronary heart disease, who have participated in a previous screening study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Quantification of coronary calcium | 2 years

SECONDARY OUTCOMES:
Determine the relationship between calcification scores and vascular reactivity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States